CLINICAL TRIAL: NCT01822353
Title: The Effect of Per Oral Immunotherapy in Severe IgE Mediated Egg, Milk and Nut Allergy in Adults
Brief Title: The Effect of Per Oral Immunotherapy in Severe IgE Mediated Egg, Milk, and Nut Allergy in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Paula Kauppi, MD, PhD, MD, PhD, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS21813030112
Record Dates: First submitted 2013-03-07; First posted 2013-04-02 (Estimated); Results first posted 2019-08-09 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Food Allergy
Keywords: food allergy; milk allergy; egg allergy; nut allergy
MeSH Terms: conditions — Food Hypersensitivity; Milk Hypersensitivity; Egg Hypersensitivity; Nut Hypersensitivity | interventions — Dietary Supplements; Milk; Egg Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Milk allergy (Experimental): Dietary supplement, milk in increasing dosages, delivered daily and orally.
  Interventions: Dietary Supplement: Dietary supplement
- Egg allergy (Experimental): Dietary supplement, egg protein given in increasing dosages, delivered daily and orally.
  Interventions: Dietary Supplement: Dietary supplement
- Nut allergy (Experimental): Dietary supplement, nut cream including nut allergens, delivered in increasing dosages, daily and orally.
  Interventions: Dietary Supplement: Dietary supplement

INTERVENTIONS:
Dietary Supplement: Dietary supplement — Milk, egg or nut oral immunotherapy
  Other Names: Milk; Egg protein; Nut cream

SUMMARY:
In Finland, the estimated prevalence of physician-diagnosed food allergy in 1-4 year old children is 9%, and the most common allergen is milk. The overall food allergy has been reported to be 3.7%. Hen's egg allergy is among the most common food allergies in childhood. In addition, it predicts later development of allergic disease such as asthma. Most of the egg and milk allergy is transient and disappears in childhood. Currently, the standard of care for food allergy includes strict allergen avoidance. However, oral immunotherapy has been under investigation in children milk, egg, and wheat allergy. Previously, induction of clinical egg tolerance has been reported with egg oral immunotherapy in children aged from 3 to 13 years. In adults, strict avoidance is still the standard care but there is also growing interest in treatment of severe food allergy with oral immunotherapy or anti-IgE.

The investigators aim to analyse the results of per oral immunotherapy treatment in severe IgE-mediated egg, milk, and nut allergy in adults.

Could severe egg, milk and nut allergy be treated with oral immunotherapy treatment in stead of total allergen avoidance and could desensitization thus be achieved?

DETAILED DESCRIPTION:
Up to 100 subjects are studied. All subjects are adults having no other severe chronic diseases. The subjects belong to four different groups:

1. 30 18-50 year olds who start per oral immunotherapy treatment in severe egg allergy.
2. 30 18-50 year olds who start per oral immunotherapy treatment in severe milk allergy.
3. 30 18-50 year olds who start per oral immunotherapy treatment in severe nut allergy.
4. 10 milk allergic 18-50 year olds that have been treated as pilot patients with milk hyposensitisation treatment.

The diagnosis of milk or egg allergy is verified with positive history, skin prick test, egg, milk and nut allergen specific IgE antibodies. In addition, food allergy is verified with an allergen specific challenge test.

Atopic subjects may have simultaneously other allergies. Intermittent mild asthma, and mild and moderate persistent asthma are tolerated and treatment with inhaled steroids and other asthma medication is allowed. Atopic subjects may have additional skin symptoms. Quality of life, anxiety and patient history data is collected by questionnaires. All patients undergo a spirometry with a bronchodilatation test, fractional exhaled nitric oxide and a methacholine challenge before and a year after oral immunotherapy. Those with test results diagnostic for asthma are treated with asthma medication before hyposensitisation treatment is started.

Exclusion criteria: adults with instable cerebrovascular or heart disease, active autoimmune disease or cancer, or use of betablocker agents. In addition, poorly controlled asthma or FEV1 < 70% are not tolerated.

In oral immunotherapy, increasing doses are given first observed, and then daily at home. If the subject does not tolerate a given dose and symptoms are mild, then that dose or the previously tolerated one is repeated, and the protocol proceeds as outlined. If the subject experiences significant symptoms, then the protocol is stopped, and the highest tolerated dose is used as the starting daily one.

ELIGIBILITY:
Inclusion Criteria:

* severe IgE-mediated milk allergy or
* severe IgE-mediated egg allergy or
* severe IgE-mediated nut allergy or
* 18-50 years

Exclusion Criteria:

* instable cerebrovascular or heart disease
* active autoimmune disease or cancer
* use of betablocker agents
* poorly controlled asthma
* FEV1 < 70% of the predicted

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mika J Mäkelä, MD, PhD, Study Director — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Milk Allergy: Dietary supplement, milk in increasing dosages, delivered daily and orally.
  Dietary supplement: Milk oral immunotherapy
- Nut Allergy: Dietary supplement, nut cream including nut allergens, delivered in increasing dosages, daily and orally.
  Dietary supplement: Nut oral immunotherapy
- Egg Allergy: Dietary supplement, egg protein given in increasing dosages, delivered daily and orally.
  Dietary supplement: Egg oral immunotherapy
Period: Overall Study
Arm/Group | Milk Allergy | Nut Allergy | Egg Allergy
Started | 10 | 9 | 4
Completed | 6 | 4 | 3
Not Completed | 4 | 5 | 1
Not completed — Adverse Event | 1 | 3 | 1
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Milk Allergy | Nut Allergy | Egg Allergy | Total
Number analyzed (Participants) | 10 | 9 | 4 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 4 | 23
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 4 | 19
  Male | 1 | 3 | 0 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Finland | 10 | 9 | 4 | 23
Allergen specific IgE [Mean (Standard Deviation); unit: kU/l] — Allergen specific IgE (casein/Arah 2 /ovomucoid) (kU/l).
  kU/l | 57.8 (60.4) | 48.8 (104.1) | 22.4 (15.5) | 47.7 (75.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of the Patients That Achieve Higher Tolerance of Allergen With Immunotherapy
Description: Number of the patients that achieve higher tolerance of allergen with immunotherapy in one year than the measured baseline allergen challenge shows.
Time Frame: One year
Measure: Number; unit: participants
Arm/Group | Milk Allergy | Nut Allergy | Egg Allergy
Number analyzed (Participants) | 10 | 9 | 4
participants | 6 | 4 | 3

2. Secondary Outcome: Effect of Therapy on Lung Function.
Description: Does hyposensitisation change lung function (do spirometry tests show difference from the baseline values (= before immunotherapy) after the immunotherapy) ?
Time Frame: One year
Measure: Mean (Standard Deviation); unit: percentage of predicted value
Arm/Group | Milk Allergy | Nut Allergy | Egg Allergy
Number analyzed (Participants) | 10 | 9 | 4
percentage of predicted value
  FEV1 (%) before OIT | 91.4 (7.4) | 96.1 (13.8) | 86.1 (8.9)
  FEV1 (%) OIT | 92.1 (6.0) | 96.3 (7.4) | 84.0 (12.1)

3. Secondary Outcome: Does Oral Immunotherapy Change Bronchial Hyperreactivity?
Description: Does bronchial hyperreactivity (measured with methacholine bronchial challenge test) show change from the baseline level after the immunotherapy?
Time Frame: One year
Population: Drop out in the number of study individuals in the methacholine measurements at one year after OIT
Measure: Mean (Standard Deviation); unit: Dose of methcholine, ug
Arm/Group | Milk Allergy | Nut Allergy | Egg Allergy
Number analyzed (Participants) | 10 | 9 | 4
Dose of methcholine, ug
  Before OIT | 531.3 (696.1) | 1303.9 (1589.0) | 691.2 (507.4)
  After OIT: number analyzed (Participants) | 1 | 1 | 4
  After OIT | 615.5 (0.0) | 2059.0 (0.0) | 973.4 (1029.1)

4. Secondary Outcome: Does the Oral Immunotherapy Have en Effect on Airway Inflammation?
Description: Does the oral immunotherapy change exhaled nitric oxide levels (measured before and after immunotherapy)
Time Frame: One year
Measure: Mean (Standard Deviation); unit: ppb
Arm/Group | Milk Allergy | Nut Allergy | Egg Allergy
Number analyzed (Participants) | 10 | 9 | 4
ppb
  Before OIT | 45.3 (36.7) | 25.7 (19.2) | 66.6 (51.3)
  After OIT | 22.5 (18.9) | 25.7 (18.1) | 66.2 (60.2)

5. Other Pre Specified Outcome: Safety of Oral Immunotherapy in Severe IgE Mediated Food Allergy in Adults.
Description: How many of the patients have side effects (categorized as mild, moderate or severe)of the hyposensitisation and how many of the patients discontinue the therapy because of side effects?
Time Frame: One year
Measure: Number; unit: Participants
Arm/Group | Milk Allergy | Nut Allergy | Egg Allergy
Number analyzed (Participants) | 10 | 9 | 4
Participants
  Mild side effects | 1 | 2 | 1
  Moderate side effects | 1 | 0 | 0
  Severe side effects | 0 | 1 | 0
  Quitting because of side effects | 1 | 2 | 1

6. Other Pre Specified Outcome: Effect of Treatment on Quality of Life
Description: Quality of life is assessed by a questionnaire before and after immunotherapy (VAS scale on worries on allergy 0-100, 0 no worries, 100 maximal worries).
Time Frame: one year
Population: Drop out in answers for quality of life at one year after OIT
Measure: Mean (Standard Deviation); unit: VAS score (mm)
Arm/Group | Milk Allergy | Nut Allergy | Egg Allergy
Number analyzed (Participants) | 10 | 9 | 4
VAS score (mm)
  Before OIT | 83.9 (15.1) | 63.5 (23.3) | 61.0 (13.0)
  After OIT: number analyzed (Participants) | 10 | 0 | 0
  After OIT | 73.0 (5.0) |  |

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Milk Allergy | Nut Allergy | Egg Allergy
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/10 | 1/9 | 0/4
Other Adverse Events (participants affected / at risk) | 8/10 | 6/9 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Milk Allergy (N=10) | Nut Allergy (N=9) | Egg Allergy (N=4)
Systemic allergic reaction (Immune system disorders) | 2 | 1 | 0 — Use of epinephrin because of allergic symptoms
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Milk Allergy (N=10) | Nut Allergy (N=9) | Egg Allergy (N=4)
Mouth and throat itching (Gastrointestinal disorders) | 8 | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2012-10-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT01822353/Prot_000.pdf
  • Statistical Analysis Plan (2012-10-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT01822353/SAP_001.pdf